CLINICAL TRIAL: NCT02498184
Title: Perioperative Acupuncture for Impacted Mandibular Third Molar Extractions - a Double Blinded Randomized Controlled Trial
Brief Title: Perioperative Acupuncture for Impacted Mandibular Third Molar Extractions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0064-15-ZIV
Record Dates: First submitted 2015-07-13; First posted 2015-07-15 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Extraction of Third Molar Teeth
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- real acupuncture (Experimental): traditional chinese acupuncture
  Interventions: Other: acupuncture
- sham acupuncture (Sham Comparator): non effective acupuncture
  Interventions: Other: acupuncture

INTERVENTIONS:
Other: acupuncture

SUMMARY:
This is a double-blinded, randomized, controlled study on the effect of perioperative acupuncture on pain after third molar extraction.

DETAILED DESCRIPTION:
Perioperative acupuncture for impacted mandibular third molar extractions - a double blinded randomized controlled trial.

The extraction of impacted third molar teeth is one of the most common surgical procedures performed by oral and maxillofacial surgeons. Post operative pain (POP) remains a significant challenge for all healthcare providers, and is a common complaint after dental and maxillofacial. NSAIDs are commonly used to treat POP and inflammation following a surgical procedure, but they are associated with unwanted side effects and can delay post operative recovery. . Third molar surgeries are associated with significant postoperative morbidity. Many clinicians have emphasized the necessity for better pain control in patients who undergo third molar surgery. Two recent systematic reviews of randomized clinical trials evaluating clinical evidence of the efficacy of acupuncture for postoperative pain control have concluded that perioperative acupuncture may be a useful adjunct for acute postoperative pain. The investigators propose a double-blinded, randomized, controlled study on the effect of perioperative acupuncture on pain in third molar surgery. Methods: 100 patients about to undergo impacted third molar extraction will be recruited. After signing an informed consent, patients will be randomized into two groups: real acupuncture and sham acupuncture. In both groups needles will be placed prior to dental treatment and will be left in place until treatment ends. Prior to treatment, all participants will fill a dental anxiety questionnaire. All patients will receive a detailed explanation regarding the dental procedure. Pre emptive etodolac 400mg will be given prior to starting the procedure. The operation will be performed under local anesthesia. Upon completion of the extraction, local lavage will be performed with physiological saline. If necessary, sutures will be placed using Rapid Vicryl 4/0. Antibiotics will not be given routinely. Patients will be advised to use Etodolac 400mg every 8 hours for the next 3 days, and to perform mouthwashes using commercially available Chlorhexidine digluconate 0.2% starting the following day. Patient follow up and data collection: Pain will be assessed using a VAS (Visual Analog Scale) by an attending nurse blinded to the randomization status, with no knowledge of acupuncture point location. VAS score will be recorded 10 minutes after the start of dental treatment and at treatment's end. Blood pressure and heart rate will be recorded during the procedure every 10 minutes. Post discharge follow up: On the day following discharge patients will be interviewed by telephone and asked to grade their general pain sensation, their ability to perform daily functions and the amount and type of analgesics they used. Inclusion criteria: Otherwise healthy adults above 18y, who are scheduled for an impacted third molar extraction, signed informed consent. Exclusion criteria: no informed consent, coagulopathy, hematological disorder, current corticosteroid therapy, known psychiatric disorder, pregnancy, immunosuppression. Data analysis: Data will be analyzed using standard statistical tests. Study location: Ziv medical center, department of maxillofacial surgery.

ELIGIBILITY:
Inclusion Criteria: Otherwise healthy adults above 18y, who are scheduled for an impacted third molar extraction, signed informed consent.

-

Exclusion Criteria:no informed consent, coagulopathy, hematological disorder, current corticosteroid therapy, known psychiatric disorder, pregnancy, immunosuppression.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
pain scale | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Ziv Medical Center, Safed, Israel